CLINICAL TRIAL: NCT03609203
Title: Improving Self-Efficacy and Resolving Inflammaging in Allogeneic Hematopoietic Cell Transplant Survivors Through Personalized Strength Programming: A Pilot Study
Brief Title: Improving Self-Efficacy, Resolving Inflammaging Allo HSCT Survivors in Personal Training
Status: Completed | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2018NTLS073; MT2018-09R (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Allogeneic HCT Survivors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: 10 Weeks of Strength Trailing; Other: Group Nutrition Discussion: week 1, week 5 and week 10
- Controls
  Interventions: Other: 10 Weeks of Strength Trailing; Other: Group Nutrition Discussion: week 1, week 5 and week 10

INTERVENTIONS:
Other: 10 Weeks of Strength Trailing — Week 1 (pre training session): self efficacy survey; 5-point frailty assessment*; diet survey; metabolic assessment; Functional status and body composition; blood and stool sample
  Week 5: self efficacy survey; Functional status and body composition
  Week 10: self efficacy survey; 5-point frailty assessment*; diet survey; metabolic assessment; Functional status and body composition; blood and stool samples
Other: Group Nutrition Discussion: week 1, week 5 and week 10 — Week 1 (pre training session): self efficacy survey; 5-point frailty assessment*; diet survey; metabolic assessment; Functional status and body composition; blood and stool sample
  Week 5: self efficacy survey; Functional status and body composition
  Week 10: self efficacy survey; 5-point frailty assessment*; diet survey; metabolic assessment; Functional status and body composition; blood and stool samples

SUMMARY:
This protocol is a pilot study of a personalized and supervised 10-week strength training program to improve self-efficacy and resolve biomarkers of inflammaging in a cohort of allogeneic hematopoietic transplant (HCT) long-term survivors versus healthy controls.

ELIGIBILITY:
Healthy Volunteers: must be the friends or relatives of the cancer patients enrolled in this study.

Inclusion Criteria:

* HCT recipients

  * Age ≥ 18 years
  * Greater than 6 months after completing systemic multiagent chemotherapy (greater than 12 months for HCT participants) at the time of enrollment. Maintenance chemotherapy is allowed
  * In remission from cancer Off immunosuppression, or on a stable immunosuppression regimen with prednisone doses ≤ 20 mg daily, with no changes planned to the immunosuppression regimen during the study period
  * Karnofsky performance status ≥ 50% (Appendix III)
  * Platelet count ≥ 50,000 without transfusions
  * Absolute neutrophil count ≥ 1
  * Willing to complete weekly strength training sessions for 10 consecutive weeks and complete all pre- and post-testing (self-efficacy survey and research blood draw)
  * Currently reside within the Minneapolis-St. Paul metro area
  * Has an adult (age ≥ 18) friend or relative who is willing to serve as an exercise partner and healthy control for the study
  * If known diabetic: Stable doses of medications to treat diabetes within 4 weeks prior to enrollment
  * Willing and able to sign voluntary written consent
* Healthy Controls

  * Age ≥ 18 years
  * Karnofsky performance status ≥ 50%
  * Willing to complete weekly strength training sessions for 10 consecutive weeks and complete all pre- and post-testing (self-efficacy survey and research blood draw)
  * Currently reside within the Minneapolis-St. Paul metro area
  * If known diabetic: Stable doses of medications to treat diabetes within 4 weeks prior to enrollment
  * Willing and able to sign voluntary written consent

Exclusion Criteria for both Cancer Survivors and Controls

* Presence of an external central venous catheter (Hickman, PICC, etc); Port-a-cath devices that are completely internal are allowed
* Use of ≥ 20+ mg prednisone daily
* Current or planned use of investigational drugs during the study period
* Myocardial infarction or stroke within 6 months
* Heart failure graded Class IV on New York Heart Association (NYHA) scale (https://manual.jointcommission.org/releases/TJC2018A/DataElem0439.html)
* Any medical condition that the consenting medical provider deems would make the participant unsafe to perform a 10-week strength training program
* Are currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A maximum of four pairs of patient/workout partners (8 subjects) should be actively participating in the 10-week group intervention on study at a time. Participants may sign consent at anytime but then begin group participation when spots become available.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Self-reported outcomes of self-efficacy | Week 10
  To quantify the changes in self-reported outcomes of self-efficacy after ten weeks of strength training in patients compared to controls.

SECONDARY OUTCOMES:
Biomarkers of inflammaging in the blood | Week 10
  To evaluate changes in biomarkers of inflammaging in the blood of HCT recipients before and after the intervention compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Shernan G Holtan, MD, Principal Investigator — Division of Hematology, Oncology and Transplantation, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States